CLINICAL TRIAL: NCT06973044
Title: Comparison Between Continuous and Intermittent Monitoring of Abnormal Respiratory and Heart Rate in Relation to Length of Stay. A Clinical Multicenter Study of Continuous Wireless Monitoring Within the NIGHTINGALE Project
Brief Title: Continuous vs Intermittent Monitoring of Respiratory and Heart Rate in Relation to Length of Stay
Acronym: CIM-LOS
Status: Completed | Type: Observational
Sponsor: Karolinska Institutet (Other)
Responsible Party: Principal Investigator, Max Bell, MD, PhD, senior lecturer, associate professor, Karolinska Institutet
Other Study IDs: Nightingale RR study
Record Dates: First submitted 2025-05-07; First posted 2025-05-15 (Actual); Last update posted 2025-05-15 (Actual); Status verified 2025-03

CONDITIONS: Perioperative Complication; Perioperative/Postoperative Complications; Surgery-Complications
MeSH Terms: conditions — Postoperative Complications

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

INTERVENTIONS:
Device: Checkpoint Cardio wireless continuous monitoring device — Continuous monitoring of respiratory rate and heart rate

SUMMARY:
Is heart rate and respiratory rate measured continuously with a new wireless sensor better as compared to standard care, with manually measured spot checks by nurses on general wards?

Does continuous monitoring detect more abnormal respiratory- and heart rate? Are abnormal values associated with increased lenght of stay?

DETAILED DESCRIPTION:
Tachypnea is not just a sign of ventilatory problems with hypoxia, but also a precursor of sepsis, metabolic acidosis and severe pain reflecting its role as an indicator of severe derangement in many body systems. A high respiratory rate has been shown to be the most reliable vital sign to predict clinical deterioration, cardiac arrest and is even associated with higher mortality rates. Despite this, it is the vital parameter most neglected; poorly documented or not recorded at all. Studies have shown that respiratory rate is measured in less than half of cases consequently jeopardizing patient safety. The lack of understanding why respiratory rate is important and its superiority to pulse oximetry in predicting clinical deterioration may be one of the reasons why it is not measured accurately.

Badawy and colleagues stated in their study "Is everyone really breathing 20 times a minute?" that respiratory rate was inaccurately recorded and had little variation in the recordings, even in patients with cardiopulmonary compromise, findings that's been supported with later studies. Respiratory rate has traditionally not been objectively measured in general wards, but instead calculated manually over 30 seconds or a minute. This could be changed by new wireless monitoring technology. A recent large study showed that continuous measured respiratory rate together with heart rate and age in a clinical deterioration model outperformed traditional early warning scores in predicting ICU admission.

The present study evaluates heart rate and respiratory rate measured continuously with a new wireless sensor as compared to standard care, with manually measured spot checks by nurses on general wards.

ELIGIBILITY:
Inclusion Criteria:

1. ≥ 18 years of age
2. planned to go through a major high-risk surgery
3. American Society of Anesthesiologists (ASA) class 2-4 due to present comorbidities
4. planned to stay in the postoperative high dependency unit for >12hours where they also would have wired continuous monitoring.

Exclusion Criteria:

1. pregnancy
2. presence of implantable defibrillator or pacemaker
3. allergy to skin adhesives

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Surgical high-risk patients, treated at Karolinska University Hospital and UMC Utrecht
Sampling Method: Probability Sample
Enrollment: 46 (Actual)
Dates: Start 2020-11-01 (Actual); Primary Completion 2021-09-30 (Actual); Study Completion 2024-12-31 (Actual)

PRIMARY OUTCOMES:
Length of stay | Within 60 days of index surgery
  Time from index surgery to hospital discharge

SECONDARY OUTCOMES:
Frequency of monitoring | Within 60 days of index surgery
  Time spent on continuous and intermittent monitoring
Abnormal respiratory rate and abnormal heart rate | Within 60 days of index surgery
  Time spent in predefined abnormal RR and HR, with continuous and intermittent monitoring

CONTACTS AND LOCATIONS:
Locations (2):
- Sweden (2):
  - Karolinska University Hospital, Stockholm
  - Karolinska Institutet, Stockholm

IPD SHARING:
Plan to Share IPD: Undecided